CLINICAL TRIAL: NCT01872715
Title: Patient Centered Outcomes in Rosacea: An Exploratory Multi-media Analysis of the Patient Experience on Oracea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10233
Record Dates: First submitted 2013-03-15; First posted 2013-06-07 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2016-01

CONDITIONS: Papulopustular Rosacea
Keywords: Papulopustular Rosacea; Oracea; anti inflammatory doxycycline
MeSH Terms: conditions — Rosacea | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oracea (Experimental): Oracea (doxycycline USP, 40mg[30mg immediate release/ 10mg delayed release beads] taken once daily in the morning on an empty stomach, one hour before meals or two hours after.
  Oral dose for 12 weeks
  Interventions: Drug: Oracea

INTERVENTIONS:
Drug: Oracea
  Other Names: doxycycline USP, 40 mg (30 mg immediate release/ 10 mg delayed release beads)

SUMMARY:
The purpose of this study is to characterize rosacea patients', being treated with Oracea, perception through visual analog scale reporting.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 25-70 years
* Diagnosis of papulopustular rosacea
* Eligible for Oracea treatment

Exclusion Criteria:

* Allergies to components of investigational product and/or hypersensitivity to tetracyclines
* Taken systemic therapy directed at improving rosacea, including antibiotics, within 30 days prior to baseline visit
* Used topical rosacea treatment within 30 days prior to baseline visit
* Have active ocular rosacea and/or blepharitis/meibomianitis requiring systemic treatment by an opthalmologist
* Previously failed to have improvement of rosacea with appropriate use of systemic tetracycline family of antibiotics
* Exposed to intense/excessive ultraviolet (UV) radiation within one week prior to baseline and/or who forsee unprotected and intense/excessive UV exposure during the course of the study
* Have planned surgical procedures during the course of the study
* Have used tetracycline antibiotics within 30 days prior to baseline visit or during study
* At risk in terms of precautions, warnings, and contraindications

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stephens & Associates Dallas Research Center, Carrollton, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oracea: Oracea (doxycycline USP, 40mg[30mg immediate release/ 10mg delayed release beads] taken once daily in the morning on an empty stomach, one hour before meals or two hours after.
  Oral dose for 12 weeks
  Oracea
Period: Overall Study
Arm/Group | Oracea
Started | 24
Completed | 20
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | Oracea
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.04 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Years since the first rosacea diagnosis [Mean (Standard Deviation); unit: years] | 5.75 (8.36)
Skin type [Number; unit: participants]
  Dry | 8
  Normal | 4
  Oily | 1
  Combination | 11
Fistzpatrick Skin Type [Number; unit: participants] — Fitzpatrick skin type is a numerical classification scale for the color of skin from Type 1 to Type VI. Skin type 1 = always burns and never tans (light, pale skin) and skin type VI = never burns, tans very easily, and is deeply pigmented (black, very dark brown to black skin).
  participants
    I | 2
    II | 15
    III | 5
    IV | 2
    V | 0
    VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Rosacea Score on the Visual Analog Scale
Description: VAS = visual analog scale, 10 cm scale in which 0 = no rosacea, 10 = worst rosacea imaginable
Time Frame: Baseline, Weeks 2, 6, and 12
Population: Intent-to-Treat (ITT) population: All subjects who were enrolled and had at least 1 posttreatment administration evaluation. This is the primary population for efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oracea
Number analyzed (Participants) | 22
units on a scale
  Baseline | 4.50 (1.81)
  Week 2 | 4.52 (1.87)
  Week 6 | 3.77 (1.93)
  Week 12 | 3.06 (2.34)

2. Secondary Outcome: Rosacea-Specific Quality of Life Index
Description: ROSACEA-SPECIFIC QUALITY OF LIFE INDEX©: average of scores to 22 questions on a 5 point scale (1 = never, 5 = all the time)
Time Frame: Baseline, Weeks 2, 6, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oracea
Number analyzed (Participants) | 22
units on a scale
  Baseline | 3.34 (0.55)
  Week 2 | 3.07 (0.56)
  Week 6 | 2.89 (0.81)
  Week 12 | 2.85 (0.86)

3. Secondary Outcome: Patient Global Assessment (PGA) of Rosacea Scores
Description: Patient Global Assessment (PGA) of Rosacea: 0 = clear, no signs or symptoms present; 1 = Near clear, 1 or 2 papules; 2 = mild, some (3 to 10) papules/pustules; 3 = moderate, moderate (11 to 19) number of papules and pustules; 4 = severe, numerous (≥ 20) papules/pustules; nodules
Time Frame: Baseline, Weeks 2, 6, and 12
Measure: Number; unit: participants
Groups:
- 0 = Clear; 1 = Near Clear; 2 = Mild; 3 = Moderate; 4 = Severe: Oracea (doxycycline USP, 40mg[30mg immediate release/ 10mg delayed release beads] taken once daily in the morning on an empty stomach, one hour before meals or two hours after; Oral dose for 12 weeks
Arm/Group | 0 = Clear | 1 = Near Clear | 2 = Mild | 3 = Moderate | 4 = Severe
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
participants
  Baseline | 0 | 1 | 17 | 4 | 0
  Week 2 | 0 | 4 | 16 | 2 | 0
  Week 6 | 0 | 10 | 11 | 1 | 0
  Week 12 | 3 | 14 | 4 | 1 | 0

4. Secondary Outcome: Patient Satisfaction Question
Description: The patient satisfaction question was answered by the subject at week 2, week 6, and week 12. The subject was asked how satisfied they were with this treatment (doxycycline MR) for rosacea.
Time Frame: Week 2, 6, and 12
Measure: Number; unit: participants
Groups:
- Very Satisfied; Satisfied; Neither Satisfied Nor Dissatisfied; Dissatisfied; Very Dissatisfied: Oracea (doxycycline USP, 40mg[30mg immediate release/ 10mg delayed release beads] taken once daily in the morning on an empty stomach, one hour before meals or two hours after; Oral dose for 12 weeks
Arm/Group | Very Satisfied | Satisfied | Neither Satisfied Nor Dissatisfied | Dissatisfied | Very Dissatisfied
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22
participants
  Week 2 | 1 | 11 | 8 | 2 | 0
  Week 6 | 4 | 7 | 8 | 2 | 1
  Week 12 | 8 | 6 | 5 | 2 | 1

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Oracea
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 7/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oracea (N=24)
Diarrhea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days